CLINICAL TRIAL: NCT03887442
Title: Phase II, Randomized Clinical Trial to Assess the Efficacy of Paclitaxel vs Paclitaxel + Cetuximab in Subjects With Recurrent and/or Metastatic Squamous Head & Neck Carcinoma After Failure of a 1º Line Chemotherapy EXTREME Type Treatment
Brief Title: Paclitaxel vs Paclitaxel + Cetuximab in Recurrent - Metastatic Head & Neck Carcinoma After Failure of a 1º Chemotherapy
Acronym: EXTAX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTCC-2009-04
Record Dates: First submitted 2011-02-11; First posted 2019-03-25 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Cetuximab; Erbitux; Paclitaxel; Extreme; Metastatic; Recurrent
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Paclitaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel (Active Comparator): Paclitaxel 80 mg/m2 may be infused, intravenously, every week.
  Interventions: Drug: Paclitaxel
- Cetuximab + Paclitaxel (Experimental): Cetuximab 250 mg/m2 and Paclitaxel 80 mg/m2, both may be infused intravenously, every week. Cetuximab will be administered prior to paclitaxel.
  Interventions: Drug: Cetuximab + Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 80 mg/m2 may be infused, intravenously, every week.
  Arms: Paclitaxel
Drug: Cetuximab + Paclitaxel — Cetuximab 250 mg/m2 and Paclitaxel 80 mg/m2, both may be infused intravenously, every week. Cetuximab will be administered prior to paclitaxel.
  Arms: Cetuximab + Paclitaxel

SUMMARY:
Treatment of recurrent and/or metastatic head and neck squamous cell carcinoma (HNSCC) after progression to first line EXTREME-type treatment in patients undergoing maintenance treatment with cetuximab.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent
2. Age ≥ 18 and < 75 y
3. ECOG (Eastern Cooperative Oncology Group)performance status: 0-1
4. Life expectancy of at least 12 weeks
5. Histological or cytological confirmation of head & neck squamous cell carcinoma with localization in larynx, oropharynx, oral cavity or hypopharynx.
6. Having received at least 2 cycles of EXTREME-type chemotherapy (cisplatin or carboplatin + fluoropyrimidines + cetuximab) and being in maintenance phase with cetuximab because of having reached CR (Complete response), PR (Partial response) or SD (Stable disease) to said treatment
7. At least one measureable lesion by CT scan or MRI
8. Adequate bone marrow, liver and kidney function, according to:

   * Hb (Hemoglobin) ≥ 9.0 g/dl
   * Platelets 100,000/mm3
   * ANC (Absolute Neutrophil Count) ≥ 1,500/mm3
   * Total bilirubin ≤ 2 times the UNL
   * SGPT/ALT and SGOT/AST ≤ 3 x UNL (Upper normal limit)
   * Alkaline phosphatase ≤ 2.5 x UNL
   * Serum creatinine ≤ 1.5 times the ULN or creatinine clearance > 50 ml/min
9. Adequate nutritional status: weight loss < 20% in relationship to usual weight or albumin ≥ 35 g/l, in the last 12 w
10. Seric calcium adjusted to albumine lower or equal to 1,25 UNL.
11. Toxicity, due to previous treatment received, resolved to grade 1, before enrolment in the study
12. Women of childbearing potential should have a (-)ve pregnancy test in serum or urine,7 d before randomization. Postmenopausal women should have remained amenorrheic for at least 12 m. Furthermore, all men as well as women who participate in this study should use effective contraceptive methods beginning with the signing of the informed consent form and up to at least 6 m after the completion of the study or of the last dose, whichever occurs first

Exclusion Criteria:

1. Treatment for recurrent and/or metastatic disease other than the EXTREME- type first line (cisplatin or carboplatin + fluoropyrimidines + cetuximab)
2. Non-measurable lesion as only evidence of disease
3. Nasopharyngeal carcinoma
4. Clinical or radiographic evidence of brain metastases
5. Having history of or presenting clinically significant cardiovascular disease, such as, but not limited to, congestive heart failure, ≥ grade II of the NYHA, severe cardiac arrhythmias that require medication, or ≥ grade II peripheral vascular disease. Furthermore, those patients who have suffered myocardial infarction or unstable angina in the year prior to the onset of the study treatment or a recent onset angina in the last 3 m will also be excluded
6. History of or current presence of grade >1 peripheral neuropathy
7. History of active neurological disease
8. History of uncontrolled convulsive episode
9. Current ≥ 2 grade infection
10. Known infection by HIV or chronic infection by HBV or HBC or presence of uncontrolled and severe intercurrent infections or other severe and uncontrolled concomitant diseases
11. History of uncontrolled diabetes, uncontrolled HBP or hepatic condition.
12. History of pulmonary fibrosis, acute pulmonary damage or interstitial pneumonia
13. Any antineoplastic treatment within the 4 w prior to the randomization period
14. History of another neoplastic disease during the last 5 y, with the exception of cured "in situ" basal cell ca.skin carcinoma, "in situ" ca.bladder, "in situ" ca.cervix and "in situ" ca.prostate
15. Known allergy or suspicion of allergy or hypersensitivity to any component of cetuximab or paclitaxel
16. Previous treatment with monoclonal antibodies or other signal transduction inhibitors or EGFR-targeted treatment (Except for previous treatment with cetuximab)
17. Known drug abuse (exception Alcoholism)
18. Any important and uncontrolled medical, psychological, psychiatric, geographic or social problem that may interfere in the participation of the subject in the study and that does not allow for adequate follow-up and compliance with the protocol and evaluation of the study results
19. Women who are pregnant or in breast-feeding period
20. Use of any investigational new drug within the 4 w prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2012-10-02 (Actual); Study Completion 2012-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Mesía, MD, Principal Investigator — Institut Català d´Oncologia-Duran i Reynals; Juan J. Grau, MD, Principal Investigator — Hospital Clinic of Barcelona; Elvira del Barco, MD, Principal Investigator — University of Salamanca; Ruth Vera, MD, Principal Investigator — Complejo Hospitalario de Navarra

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out in 10 academic medical centers in Spain. First patient in was on 16-February-2011 and the study was closed (last patient in) on 02-October-2012.
Period: Overall Study
Arm/Group | Paclitaxel | Cetuximab + Paclitaxel
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel | Cetuximab + Paclitaxel | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.16 (7.25) | 58.48 (8.76) | 60.96 (8.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The primary endpoint was to select the most effective treatment arm based on the progression-free survival (PFS) reached in each treatment arm. This was defined as the time elapsed from inclusion in the study until the date when disease progression or death (for any cause) was documented.
Time Frame: Through study completion. The study was prematurely closed at 19 months due to lack of accrual. The primary endopoint was not analyzed.
Population: Only 17 patients out of a planned protocol number of 80 were recruited to the study, owing to premature closure of the study. Two of those patients did not meet some of the inclusion and/or exclusion criteria. Database lock: 3 June 2013. There were insufficient numbers of patients to be able to analyse the efficacy endpoints.
  The possible discrepancies that were pending resolution have been closed as "Premature closure of the study. Deviation DN13/024".
  .
Arm/Group | Paclitaxel | Cetuximab + Paclitaxel
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival
Description: Calculate overall survival (OS) in both arms
Time Frame: Through study completion. The study was prematurely closed at 19 months due to lack of accrual. The secondary endopoint was not analyzed.
Population: Only 17 patients out of a planned protocol number of 80 were recruited to the study, owing to premature closure of the study (Database lock: 3 June 2013). There were insufficient numbers of patients to be able to analyse the secondary endpoints.
  The possible discrepancies that were pending resolution have been closed as "Premature closure of the study. Deviation DN13/024".
Arm/Group | Paclitaxel | Cetuximab + Paclitaxel
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Objective Response
Description: Calculate the percentage of objective responses (OR), following the new RECIST criteria, obtained in both arms
Time Frame: Through study completion. The study was prematurely closed at 19 months due to lack of accrual. Neither the primary nor the secondary endopoints were analyzed.
Population: Only 17 patients out of a planned protocol number of 80 were recruited to the study, owing to premature closure of the study. Two of those patients did not meet some of the inclusion and/or exclusion criteria. Database lock: 3 June 2013. There were insufficient numbers of patients to be able to analyse the primary and secondary endpoints of the study
Arm/Group | Paclitaxel | Cetuximab + Paclitaxel
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Participants With Adverse Events
Description: To perform a descriptive analysis of the adverse events observed in the patients included in the study. Further analysis could not be performed due to early closure of this study due to lack of accrual. Adverse events were registered from study entry until 60 days after receiving the last dose of study drug.
Time Frame: The duration of the study (Nineteen months) and until the last patient included completed one year of follow up / died or was lost to FU. Adverse events were registered from study entry until 60 days after receiving the last dose of study drug.
Population: This safety analysis includes all 17 patients (Database lock: 3 June 2013). There were insufficient numbers of patients to be able to analyse the efficacy endpoints.
  The possible discrepancies that were pending resolution have been closed as "Premature closure of the study. Deviation DN13/024".
Measure: Number; unit: participants
Arm/Group | Paclitaxel | Cetuximab + Paclitaxel
Number analyzed (Participants) | 9 | 8
participants | 9 | 8

5. Secondary Outcome: Treatment Compliance
Description: Evaluate treatment compliance rate in both treatment arms, in order to analyze it, the dose intensity would be calculated as the quantity of each of the administered study drugs per unit of time (mg/m2/week) regardless of the treatment arm. To analyze the relative dose intensity, the dose of each administered drug will be divided per a unit of time and the planned quantity of each drug according to the doses described in the protocol.
Time Frame: 3 years
Population: Only 17 patients out of a planned protocol number of 80 were recruited to the study, owing to premature closure of the study (Database lock: 3 June 2013). There were insufficient numbers of patients to be able to analyse the primary and secondary endpoints.
  The possible discrepancies that were pending resolution have been closed as "Premature closure of the study. Deviation DN13/024".
Arm/Group | Cetuximab + Paclitaxel | Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected across the duration of study treatment. This was during the 19 months the study was open until 60 days after the last patient being treated received the last dose of study drug.
Arm/Group | Paclitaxel | Cetuximab + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 6/9 | 4/8
Serious Adverse Events (participants affected / at risk) | 4/9 | 4/8
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=9) | Cetuximab + Paclitaxel (N=8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fracture of humerus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (2)
Pneumococcal pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=9) | Cetuximab + Paclitaxel (N=8)
Edema (General disorders) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6)
Peripheral neuropathy (Nervous system disorders) | 2 (6) | 1 (4)
Asthenia (General disorders) | 5 (8) | 5 (16)
Post-surgical wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Pain in an extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Naso-pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (3)
Mucosal inflammation (General disorders) | 3 (4) | 6 (14)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (6) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypoesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (5) | 0 (0)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Tracheal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palmoplantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Peripheral edema (General disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (7) | 2 (2)
Xerosis (General disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Loss of hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Face swelling (General disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Mouth bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bad breath (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear ache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (4) | 1 (3)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Sensory peripheral neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (4) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loss of appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervicalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Excessive tearing (Eye disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (3)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (6)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Tracheal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Swollen eyelids (Eye disorders) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mouth pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teeth deterioration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Decline in general physical status (General disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mass in neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
After 19 mos. the study was prematurely closed due to lack of accrual, only 17 pts were included. It was not possible to analyze the 1ry nor the 2ry endpoints of the study. A safety analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No